CLINICAL TRIAL: NCT07341477
Title: Microbiome and Health-related Effects of a Dietary Supplement in Infants: a Double-blind, Randomized, Placebo-controlled Nutritional Study.
Brief Title: Efficacy of a Dietary Supplement in Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2406INF
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Infants
Keywords: Dietary Supplement
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled nutritional study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unique (individual) coding of the study products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental)
  Interventions: Dietary Supplement: Experimental Group
- Control Group (CG) (Placebo Comparator)
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Dietary Supplement: Experimental Group — Dietary supplement in powder form
  Arms: Experimental Group (EG)
Other: Control Group (CG) — Placebo dietary supplement in powder form
  Arms: Control Group (CG)

SUMMARY:
This is a double-blind, randomized, placebo-controlled nutritional study of healthy term infants. The primary objective of the trial is to demonstrate a favorable change in fecal microbiome composition in infants receiving a dietary supplement compared to infants receiving a placebo supplement.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled nutritional study of healthy term infants, consisting of 2 randomized parallel arms: experimental group (EG) receiving a dietary supplement and a control group (CG) receiving a placebo supplement.

The population under investigation is healthy infants aged 5 months +/- 1 week at the time of clinic visit 1.

The planned sample size for this study is 172 infants (86 per study group). Each investigational product (EG and CG) will be provided in powder form and packaged in single dose stick packs. The powder will be dissolved in lukewarm formula or body temperature breastmilk and fed orally to the infants using a provided infant feeding beaker.

The primary objective of the trial is to demonstrate a favorable change in fecal microbiome composition in infants receiving a dietary supplement compared to infants receiving a placebo supplement from enrolment until 5 months of intervention.

In addition, fecal metabolic biomarkers, gastrointestinal (GI) related outcomes, blood markers of immune health, fecal markers of gut and immune health, bone quality, other anthropometric measurements, dietary pattern and infant illness and infection outcomes will be assessed/measured.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from at least one parent (or legally acceptable representative [LAR])
2. Parent(s) / LAR(s) must be able to provide evidence of parental authority and identity
3. Parent(s) / LAR(s) must understand the informed consent form and other study documents
4. Parent(s) / LAR(s) are willing and able to comply with scheduled visits and the requirements of the study protocol including infant blood collection
5. Parent(s) / LAR(s) can be contacted directly by telephone throughout the study
6. Parent(s) / LAR(s) must be able to temporarily store stool samples in a household freezer
7. Parent(s) / LAR(s) of formula-fed infants (either exclusively or mixed-fed) must have previously and independently decided to use formula and their infant must be consuming and tolerating a standard cow's milk infant formula not containing probiotics at the time of enrollment
8. Infant must be healthy based on medical history and physical examination
9. Infant full-term gestational birth (born 37 weeks, 0 days through 41 weeks, 6 days)
10. Infant age 5 months ± 1 week (date of birth = day 0) at time of clinic visit 1
11. Infant birth weight is appropriate for gestational age (i.e., ≥ 2500 and ≤ 4500 grams)

Exclusion Criteria:

1. Infants with conditions requiring specific infant feeding regimens other than those specified in the protocol
2. Infants receiving solid foods or liquids other than breastmilk or infant formula within 4 weeks prior to enrollment
3. Infants who have a medical condition or medical history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation)
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis)
   3. Immunocompromised infants and those who have a central venous catheter
   4. History of admission to the Neonatal Intensive Care Unit, except for admission for jaundice phototherapy.
   5. Known or suspected allergy to milk (including lactose) or soy
   6. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgement of the investigator, would make the infant inappropriate for entry into the study.
4. Infants who are currently receiving or who have received any probiotic supplements or any infant formula containing probiotics prior to enrollment
5. Infants who are currently receiving or who have previously received any of the following medication(s) or supplement(s) which are known or suspected to affect fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes), stool characteristics (e.g., glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose), growth (e.g. insulin or growth hormone), microbiome-related endpoints (e.g., prebiotic supplements, antibiotic usage within the past 4 weeks [not including topical or ophthalmic applications]), or gastric acid secretion.
6. Infants whose parent(s) / LAR(s) have not reached the legal age of majority (18 years old)
7. Infants who are currently or who previously participated in another interventional clinical study
8. Parent(s) / LAR(s) with family or hierarchical relationships with the research team members

Ages: 19 Weeks to 21 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Probiotic abundance | At 5 months (V4) of intervention
  Fecal probiotic abundance

SECONDARY OUTCOMES:
Fecal metabolic biomarker | At baseline (V1), 3 months (V3), and 5 months (V4) of intervention.
  To assess changes in key fecal metabolic biomarkers such as fecal water-soluble vitamins, fecal organic acids, and other fecal metabolites.
Growth parameter: Weight | At baseline (V1), 1 month (V2), 3 months (V3), and 5 months (V4) of intervention.
  Weight in grams and corresponding weight-for-age Z-score according to WHO growth standards
Growth parameter: Length | At baseline (V1), 1 month (V2), 3 months (V3) and 5 months (V4) of intervention.
  Length in cm and corresponding weight-for-age Z-score according to WHO growth standards
Growth parameter: Head circumference | At baseline (V1), 1 month (V2), 3 months (V3) and 5 months (V4) of intervention.
  Head circumference in cm and corresponding head circumference-for-age Z-score according to WHO growth standards
GI-related Behavior: Infant Gastrointestinal Symptom Questionnaire (IGSQ) | At baseline (V1), 1 month (V2), 3 months (V3) and 5 months (V4) of intervention.
  The questionnaire is composed of 13 questions, categorized into 5 symptom domains of stooling, vomiting/spitting-up, crying, fussiness, and flatulence. The total score can range from 13 to 65 with lower scores indicating lower GI symptom burden.
GI-related behavior: Stool frequency | 1-day retrospective (V1) and 3-day prospective (V2, V3 and V4) of intervention
  Stool frequency recorded via the GI Symptom and Behavior Diary
GI-related behavior: Stool consistency | 1-day retrospective (V1) and 3-day prospective (V2, V3 and V4) of intervention
  Stool consistency recorded on a 5-point scale (1: watery, 5: hard) via the GI Symptom and Behavior Diary
GI-related behavior: Crying and sleeping | 1-day retrospective (V1) and 3-day prospective (V2, V3 and V4) of intervention
  Crying and sleeping time via the GI Symptom and Behavior Diary
Fecal microbiota | At baseline (V1), 1 month (V2), 3 months (V3), and 5 months (V4) of intervention.
  Overall fecal microbiota composition, diversity, and function.
Bone quality | At baseline (V1), 3 months (V3), and 5 months (V4) of intervention.
  Tibia bone transmission time and speed of sound. Tibia length assessed using a measuring tape.
Dietary intake: Food record | 3 consecutive days prior to study visit 3 (age 8 months) and visit 4 (age 10 months)
  Dietary intake using a 3-day food record completed at home
Dietary intake: Complementary foods | Questionnaire to be completed prospectively starting at age 6 months
  Exact timing of the introduction of different types of complementary foods assessed using the Complementary Food Questionnaire
Dietary intake: Formula Composition | At baseline (V1), 1 month (V2), 3 months (V3), and 5 months (V4) of intervention.
  Key aspects of formula composition assessed using a questionnaire at each study visit for formula-fed infants (exclusively or mixed-fed).
Fecal markers of gut and immune health: Formula-fed infants only | At 1 month (V2), 3 months (V3), and 5 months (V4) of intervention in exclusively formula-fed infants only.
  Fecal markers of gut and immune health such as total secretory IgA (sIgA)
Fecal markers of gut and immune health: All infants | At baseline (V1), 1 month (V2), 3 months (V3), and 5 months (V4) of intervention in all infants.
  Fecal markers of gut and immune health such as fecal pH, fecal calprotectin, fecal α-1-antitrypsin, oral vaccine-specific fecal antibodies.
Blood biomarkers | At baseline (V1), 3 months (V3), and 5 months (V4) of intervention.
  Blood biomarkers such as immunotyping, plasma immune proteomics, metabolic and anabolic biomarkers, plasma metabolomics, vaccine-specific antibodies, plasma short-chain fatty acids.
Neurodevelopment: National Institute of Health (NIH) Baby Toolbox | At 5 months (V4) of intervention
  To assess different aspects of infant neurodevelopment
Neurodevelopment: Heart rate variability | Assessed for 24 hours at home after baseline (V1), 3 months (V3), and 5 months (V4) of intervention.
  Heart rate variability will be assessed using a simple, non-invasive sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mitzi Trinidad-Aseron, Principal Investigator — University of Perpetual Help Dalta Medical Center, Philippines; Dr. Maria Josefa Nantes, Principal Investigator — Silang Specialists Medical Center, Philippines

IPD SHARING:
Plan to Share IPD: No